CLINICAL TRIAL: NCT07343063
Title: Evaluation of Anterior Restorations
Brief Title: Evaluation of the Clinical Performance of Different Composite Materials in Class III and IV Restorations.
Status: Recruiting | Type: Observational
Sponsor: Recep Tayyip Erdogan University (Other)
Responsible Party: Principal Investigator, Muhammet Karadaş, Clinical Professor, Recep Tayyip Erdogan University
Other Study IDs: RTEUDHFMKARADAS006
Record Dates: First submitted 2026-01-06; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Dentin Caries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Composite materials — Restorations

SUMMARY:
In this study, a universal adhesive was used with different adhesive techniques (self-etch and total-etch modes) and evaluated for 18 months in three different types of composite material class III and class IV restorations according to the FDI criteria. The hypotheses tested in this study are: (1) clinical success will not differ between different composite materials and (2) clinical outcomes will not differ between different application modes of the universal adhesive.

ELIGIBILITY:
Inclusion Criteria:

* Good general health
* No heart disease,
* No diabetes
* No systemic diseases such as hypertension

Exclusion Criteria:

* Individuals with advanced periodontitis and associated postoperative sensitivity
* Pregnant and breastfeeding women
* Individuals undergoing orthodontic treatment and using appliances
* Individuals with direct pulp capping
* Individuals with bruxism

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All restorations to be evaluated in this study were performed at the Department of Restorative Dentistry, Faculty of Dentistry, Recep Tayyip Erdoğan University. Participants who received routine dental treatment at the university's dental clinic and whose records were kept will be included in the research.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-05-16 (Actual); Primary Completion 2027-01-16 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
FDI criteria | 2 years
  very good, good, poor, very poor

CONTACTS AND LOCATIONS:
Locations (1):
- Muhammet Karadaş, Merkez, Rize Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No